CLINICAL TRIAL: NCT00994916
Title: Treatment of Lambert-Eaton Syndrome With 3,4 Diaminopyridine
Status: No longer available | Type: Expanded Access
Sponsor: David Lacomis, MD (Other)
Collaborators: Jacobus Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, David Lacomis, MD, Professor of Neurology and Pathology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: IRB0410047
Record Dates: First submitted 2009-10-08; First posted 2009-10-14 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Lambert-Eaton Myasthenic Syndrome
Keywords: Lambert-Eaton myasthenic syndrome; 3,4 diaminopyridine
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome | interventions — Amifampridine

INTERVENTIONS:
Drug: 3,4 diaminopyridine — 3,4 diaminopyridine up to 80 mg daily in divided doses

SUMMARY:
The purpose of the study is to provide expanded access (compassionate use) of 3,4 diaminopyridine to patients with Lambert-Eaton myasthenic syndrome (LEMS).

DETAILED DESCRIPTION:
Up to 15 patients over the age of 18 years with a diagnosis of LEMS are eligible to enroll if they are medically stable. They may receive 3,4 diaminopyridine in addition to other treatments and standard of care investigations for LEMS under supervision of the primary investigator. Safety laboratory studies and EKGs will be obtained.

The study has been approved by the University of Pittsburgh IRB. There is a local Data-Safety Monitoring Board.

The investigator has a hold on enrolling new subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of LEMS
2. Over 18 years old
3. Medically stable
4. If female and premenopausal, have a negative urine pregnancy test prior to starting the 3,4 DAP, and, if premenopausal, be willing to practice an effective form of birth control such as "double-barrier contraception" during the study

Exclusion Criteria:

1. Known sensitivity to 3,4 DAP
2. History of past or current seizures
3. History of severe asthma
4. Believed by the investigator to be unable to comply with the protocol
5. Unable to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult